CLINICAL TRIAL: NCT05279833
Title: SLR/NMA of Multaq® vs Sotalol to Assess for Safety in Patients With Atrial Fibrillation (AFib)
Brief Title: Systematic Review and Meta-Analysis of Multaq® for Safety in Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: CSA0010
Record Dates: First submitted 2022-02-17; First posted 2022-03-15 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Dronedarone; Sotalol

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: dronedarone — Pharmaceutical form is tablet and route of administration is oral
  Other Names: Multaq®
Drug: sotalol — Pharmaceutical form is tablet and route of administration is oral
  Other Names: BETAPACE®

SUMMARY:
A systematic literature review (SLR) will be conducted to understand the landscape of evidence on the relative safety and effectiveness/efficacy of dronedarone compared to sotalol in patients with AFib within interventional clinical trials and observational studies.

ELIGIBILITY:
Inclusion Criteria:

Following eligibility criteria are defined to select relevant studies from the literature

* Adults with Atrial Fibrillation(AFib) (non-permanent, including paroxysmal or persistent, long-standing persistent AFib [over 12 months]))
* Participants have received either Dronedarone or Sotalol
* controlled clinical trials or comparative observational studies( prospective/retrospective cohort, case-control studies, population-based studies or registry based studies

Exclusion Criteria:

Exclusion criteria for potential participants are:

* Children/adolescents
* Permanent atrial fibrillation (AFib)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with AFib (non-permanent, including paroxysmal or persistent, long-standing persistent AFib [over 12 months])
Sampling Method: Non-Probability Sample
Enrollment: 87810 (Actual)
Dates: Start 2021-09-24 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with Cardiovascular (CV) hospitalization | As reported in studies included in the systematic review up to 10 years
  CV hospitalization is defined as composite of heart failure hospitalization, AFib hospitalization, MI, and stroke
Number of participants with ventricular proarrhythmia | As reported in studies included in the systematic review up to 10 years
Number of all-cause mortality events | As reported in studies included in the systematic review up to 10 years
Number of cardiovascular mortality events | As reported in studies included in the systematic review up to 10 years
  includes arrhythmia-related mortality
Number of participants with atrial fibrillation (AFib) recurrence | As reported in studies included in the systematic review up to 10 years

SECONDARY OUTCOMES:
Number of participants with myocardial infarction | As reported in studies included in the systematic review up to 10 years
Number of participants with stroke | As reported in studies included in the systematic review up to 10 years
Number of participants with heart failure hospitalization | As reported in studies included in the systematic review up to 10 years
Number of participants with AFib hospitalization | As reported in studies included in the systematic review up to 10 years
Number of participants with conduction disorders | As reported in studies included in the systematic review up to 10 years
  Atrioventricular block (2nd or 3rd degree) or Requirement of pacemaker implants

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences and Operations, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, France, Chilly-Mazarin, France

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Result] Singh JP, Blomstrom-Lundqvist C, Turakhia MP, Camm AJ, Fazeli MS, Kreidieh B, Crotty C, Kowey PR. Dronedarone versus sotalol in patients with atrial fibrillation: A systematic literature review and network meta-analysis. Clin Cardiol. 2023 Jun;46(6):589-597. doi: 10.1002/clc.24011. Epub 2023 Apr 6. PMID 37025083